CLINICAL TRIAL: NCT02007863
Title: Treatment Protocol: Umbilical Cord Blood (UCB) Transplantation in Pediatric Patients With High Risk Leukemia and Myelodysplasia Using Conditioning Regimen Without Radiation
Brief Title: Umbilical Cord Blood (UCB) Transplantation in Pediatric Patients With High Risk Leukemia and Myelodysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Martin Andreansky, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080774
Record Dates: First submitted 2013-12-03; First posted 2013-12-11 (Estimated); Results first posted 2015-12-28 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-11

CONDITIONS: Leukemia; Myelodysplasia; Acute Lymphocytic Leukemia; Acute Myelogenous Leukemia
Keywords: Leukemia; Myelodysplasia; Acute lymphocytic leukemia; ALL; Acute myelogenous leukemia; AML; Pediatric
MeSH Terms: conditions — Leukemia; Anemia, Refractory, with Excess of Blasts; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — fludarabine; fludarabine phosphate; Busulfan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical Cord Blood + Chemotherapy (Experimental): Umbilical Cord Blood transfusion + Chemotherapy (Fludarabine + Busulfan + Melphalan)
  Interventions: Procedure: Umbilical Cord Blood Transfusion; Drug: Fludarabine; Drug: Busulfan; Drug: Melphalan

INTERVENTIONS:
Procedure: Umbilical Cord Blood Transfusion — Following the administration of the preparative therapy, all subjects will undergo UCB transplantation. Umbilical Cord Blood Transfusion will occur on Day 0
  Other Names: UCB
Drug: Fludarabine — Fludarabine 25 mg/m2/day will be administered over 30-60 minutes intravenous infusion on Days -13 through -9 for a total of 5 doses. Fludarabine will not be dose adjusted for body weight.
  Other Names: Fludara
Drug: Busulfan — Busulfan IV (Busulfex) will be administered IV every 6 hours on days -8 through -5 for a total of 16 doses. Seizure prophylaxis prior to first dose of busulfan till Day -3 will be administered.
  Other Names: Busulfex
Drug: Melphalan — Melphalan 45 mg/m2/day will be administered over 60 minutes intravenous infusion on Days -4 through -2 for a total of 3 doses.
  Other Names: Alkeran

SUMMARY:
Unrelated Cord Blood (UCB) transplant in children is a viable stem cell transplant modality for patients with leukemia and myelodysplasia. UCB is now considered "Standard Of Care" in cases where a suitable living bone marrow donor is not available. The survival of UCB is similar to Matched Unrelated Marrow Transplant. This study is considered "Research" since UCB is not a licensed product and requires investigational new drug (IND). THERE ARE NO SPECIFIC RESEARCH QUESTIONS IN THIS PROTOCOL. This protocol merely provides UCB as a stem cell treatment modality to pediatric patients who may require it after a conditioning regimen that excludes Total Body Irradiation.

DETAILED DESCRIPTION:
The preparative regimen will consist of:

* Fludarabine: 25 mg/m2/day IV x 5 doses on Days -13, to -9
* Busulfan 1mg/kg IV every 6 hrs x 16 doses on Days -8 to -5
* Melphalan 45 mg/m2/day IV x 3 doses on days -4 to -2
* ATGAM 30mg/kg/day x 3 doses on Days -3 to -1
* Day 0 will be the day of the UCB Transplant
* The graft-versus-host-disease (GVHD) prophylaxis will be Cyclosporin A to maintain level 200-400 beginning on Day -3, through 200-400. Solumedrol at 1mg/kg/day on Day 1 until D+4, then solumedrol 2mg/kg/day until Day +19 or till absolute neutrophil count (ANC) reaches 500/mm2, then taper by 0.2 mg/kg/week.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be up to 21 years of age
* Patients cannot receive total body irradiation (TBI) because of:

  * Young age - < 2 years at diagnosis of leukemia resulting in an age < 4 years at transplantation (due to risk of severe growth retardation and brain damage).
  * Inability to tolerate TBI because of prior radiation or organ toxicity.
  * Refractory/multiply relapsed leukemia, for which a traditional TBI/cyclophosphamide regimen would unlikely lead to a successful outcome.
* Patients must have a partially human leukocyte antigen (HLA)-matched UCB unit. Unit must be HLA-matched minimally at 4 of 6 HLA-A and B (at intermediate resolution by molecular typing) and DRB1 (at high resolution by molecular typing) loci with the patient. The unit must deliver a pre-cryopreserved nucleated cell dose of at least 2.5 x 10^7 per kilogram.
* Acute myelogenous leukemia (AML) at the following stages:

  * High risk first complete remission (CR1), defined as:

    * Having preceding myelodysplasia (MDS)
    * High risk cytogenetics (High-risk cytogenetics: del (5q) -5, -7, abn (3q), t (6;9) complex karyotype (>= 5 abnormalities)
    * Requiring > 2 cycles chemotherapy to obtain CR;
  * Second or greater CR.
  * First relapse with < 25% blasts in bone marrow.
* Patients with therapy-related AML whose prior malignancy has been in remission for at least 12 months.
* Acute lymphocytic leukemia (ALL) at the following stages:
* High risk first remission, defined as:

  1. Ph+ ALL; or,
  2. Myeloid/lymphoid leukemia (MLL) rearrangement with slow early response [defined as having M2 (5-25% blasts) or M3 (>25% blasts on bone marrow examination on Day 14 of induction therapy)]; or,
  3. Hypodiploidy (< 44 chromosomes or DNA index < 0.81); or,
  4. End of induction M3 bone marrow; or,
  5. End of induction M2 with M2-3 at Day 42.
* High risk second remission, defined as:

  1. Bone marrow relapse < 36 months from induction; or,
  2. T-lineage relapse at any time; or,
  3. Very early isolated central nervous system (CNS) relapse (6 months from diagnosis); or,
  4. Slow reinduction (M2-3 at Day 28) after relapse at any time.
* Any third or subsequent CR.
* Biphenotypic or undifferentiated leukemia in any CR or if in 1st relapse must have < 25% blasts in bone marrow (BM).
* MDS at any stage.
* Chronic myelogenous leukemia (CML) in chronic or accelerated phase.
* All patients with evidence of CNS leukemia must be treated and be in CNS CR to be eligible for study.
* Patients ≥ 16 years old must have a Karnofsky score ≥ 70% and patients < 16 years old must have a Lansky score ≥ 70%.
* Signed informed consent.
* Patients with adequate physical function as measured by:

  1. Cardiac: Left ventricular ejection fraction at rest must be > 40%, or shortening fraction > 26%
  2. Hepatic: Bilirubin ≤ 2.5 mg/dL; and alanine transaminase (ALT), aspartate transaminase (AST) and Alkaline Phosphatase ≤ 5 x upper limit of normal (ULN)
  3. Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function (creatinine clearance or GFR) > 70 mL/min/1.73 m2.
  4. Pulmonary: Diffusing capacity of the lungs for carbon monoxide (DLCO), Forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC) (diffusion capacity) > 50% of predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then O2 saturation > 92% of room air.

Exclusion Criteria:

* Pregnant (B-positive HCG) or breastfeeding.
* Evidence of HIV infection or HIV positive serology.
* Current uncontrolled bacterial, viral or fungal infection (currently taking medication and progression of clinical symptoms).
* Autologous transplant < 6 months prior to enrollment.
* Prior autologous transplant for the disease for which the UCB transplant will be performed.
* Allogeneic hematopoietic stem cell transplant < 6 months prior to enrollment.
* Active malignancy other than the one for which the UCB transplant is being performed within 12 months of enrollment
* Active CNS leukemia.
* Requirement of supplemental oxygen.
* HLA-matched related donor able to donate.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2008-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Andreasky, MD, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Umbilical Cord Blood + Chemotherapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Umbilical Cord Blood + Chemotherapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Successful Unrelated Cord Blood (UCB) Transplants
Description: The number of patients who received successful UCB transplants as evidenced by absolute neutrophil recovery.
Time Frame: 2 Years
Population: THERE ARE NO SPECIFIC RESEARCH QUESTIONS IN THIS PROTOCOL. This protocol merely provides UCB as a stem cell treatment modality to pediatric patients who may require it after a conditioning regimen that excludes Total Body Irradiation.Unrelated Cord Blood (UCB) transplant
Measure: Number; unit: participants
Arm/Group | Umbilical Cord Blood + Chemotherapy
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Arm/Group | Umbilical Cord Blood + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
THERE ARE NO SPECIFIC RESEARCH QUESTIONS IN THIS PROTOCOL. This protocol merely provides UCB as a stem cell treatment modality to pediatric patients who may require it after a conditioning regimen that excludes Total Body Irradiation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes